CLINICAL TRIAL: NCT04321447
Title: Clinical Practice Guideline on the Prevention and Management of Neonatal Extravasation Injury
Brief Title: Clinical Practice Guideline for Neonatal Extravasation Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Christian Hospital (Other)
Responsible Party: Principal Investigator, CHAN Kam Ming, Nurse Consultant, United Christian Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CPGneonatalextravasation
Record Dates: First submitted 2020-03-20; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Extravasation Injury
Keywords: Intravenous nursing; Newborn infant; Neonatal intensive care units; Evidence-based professional practice

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical practice guideline (CPG) group (Experimental): Implementation of an evidence-based clinical practice guideline and delivery of an educational programme
  Interventions: Other: Clinical practice guideline for prevention and management of extravasation injury
- Usual care group (No Intervention): Usual care

INTERVENTIONS:
Other: Clinical practice guideline for prevention and management of extravasation injury — Implementation of an evidence-based clinical practice guideline and delivery of an educational programme for nurses
  Arms: Clinical practice guideline (CPG) group

SUMMARY:
This study is aimed to evaluate the effectiveness of an evidence-based clinical practice guideline in the prevention and management of neonatal extravasation injury, and to examine the change in nurses' knowledge of and adherence to the guideline.

DETAILED DESCRIPTION:
A study with controlled before-and-after design was conducted. The clinical practice guideline was developed and a multifaceted educational program was delivered for nurses. Neonatal outcomes were collected at baseline and after completion of the intervention. The changes in nurses' level of knowledge and adherence to the guideline were also measured.

ELIGIBILITY:
Inclusion Criteria:

* Neonates who were admitted for intravenous medication or infusion therapy, and
* Neonates whose parents were equal to or over 18 years old and able to communicate in Chinese or English.

Exclusion Criteria:

* Neonates who were born with congenital dermatological problems such as ichthyosis and epidermolysis bullosa.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 213 (Actual)
Dates: Start 2015-11-14 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2017-08-29 (Actual)

PRIMARY OUTCOMES:
Change in rate of peripheral intravenous extravasation | Change from Baseline rate at one month
  The number of the incidents divided by the total number of catheter days and multiplied by 1,000
Change in rate of extravasation from a central line | Change from Baseline rate at one month
  The number of the incidents divided by the total number of catheter days and multiplied by 1,000

SECONDARY OUTCOMES:
Change in nurses' level of knowledge | Change from Baseline Knowledge level at six months
  The Neonatal Extravasation Knowledge Test
Change in nurses' adherence to clinical practice guidelines | Change from Baseline Adherence level at six months
  A 27-item audit tool

CONTACTS AND LOCATIONS:
Overall Officials: Kam Ming Chan, Principal Investigator — United Christian Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan KM, Chau JPC, Choi KC, Fung GPG, Lui WW, Chan MSY, Lo SHS. Clinical practice guideline on the prevention and management of neonatal extravasation injury: a before-and-after study design. BMC Pediatr. 2020 Sep 23;20(1):445. doi: 10.1186/s12887-020-02346-9. PMID 32967637